CLINICAL TRIAL: NCT05850468
Title: Assistant Professor of Anesthesia, Intensive Care and Pain Management
Brief Title: Effectiveness of Combining Erector Spinea Block With Non Opioid Infusions as Opioid Free Anesthesia in Spine Surgeries.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS81/2023
Record Dates: First submitted 2023-03-18; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-03

CONDITIONS: Opioid Use; Spine Fusion
Keywords: multimodal analgesia, regional blocks, spine surgeries
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- traditinal balanced anesthesia (Active Comparator): fentanyl infusion after general anesthesia and erector spinea block
  Interventions: Drug: fentanyl infusion after general anesthesia and erector spinea block
- opioid free anesthesia (Experimental): lidocaine and dextometidine infusion after general anesthesia and erector spinea block
  Interventions: Drug: lidocaine 2% and dextometometidine infusion after general anesthesia and erector spinea block

INTERVENTIONS:
Drug: fentanyl infusion after general anesthesia and erector spinea block — intraoperative opioid infusion in active comparative group
  Other Names: opioid infusion
  Arms: traditinal balanced anesthesia
Drug: lidocaine 2% and dextometometidine infusion after general anesthesia and erector spinea block — intraoperative non opioid infusion in experimental group
  Other Names: lidocaine 2% and precedex infusion
  Arms: opioid free anesthesia

SUMMARY:
opioid free anesthesia consists of combination of pharmacological and non pharmacological modalities that target different pathways of pain mechanism. combining myofascial plane blocks with infusion of adjuvants such as lidocaine or dexmedetomidine can offer equivalent intraoperative hemodynamic stability compared to that of opioid with better pain control postoperatively. this study will investigate the efficacy of combined erector spina block with lidocaine and dexmedetomidine infusion as opioid sparing anesthesia in spine surgeries

DETAILED DESCRIPTION:
patients who will undergo spine surgery will be allocated into two groups. after general anesthesia, bilateral erector spine block will be applied in both groups. group A will have intraoperative fentanyl infusion and group B will have lidocaine and dexmedetomidine infusion in 50 ml syringe till end of surgery

ELIGIBILITY:
Inclusion Criteria:

- spine surgery ASAI,II

Exclusion Criteria:

* revision surgery hypotension bradycardia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
number of patients (percentage) having intraoperative systolic hypertension | during operation(intraoperatively)
  blood pressure more than 160 mmhg
number of patients(percentage) having tachycardia | during operation(intraoperatively)
  heart rate more than 100 beat /minute

SECONDARY OUTCOMES:
VAS score | every 30 minutes for 2 hours postoperatively
  score from 0 to 10, 0 is no pain and 10 the worst pain
incidence of bradycardia | intraoperatively
  heart rate less than 45 beat per minute

CONTACTS AND LOCATIONS:
Overall Officials: sanaa wasfy, professor, Principal Investigator — assistant professor of anesthesia
Locations (1):
- Ainshams hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowland M, Thomson PD, Guichard A, Melmon KL. Disposition kinetics of lidocaine in normal subjects. Ann N Y Acad Sci. 1971 Jul 6;179:383-98. doi: 10.1111/j.1749-6632.1971.tb46915.x. No abstract available. PMID 5285383